CLINICAL TRIAL: NCT06241391
Title: Role of Ga-68 Prostate Specific Membrane Antigen PET/CT in Detection of Recurrence in Patients With Gliomas
Brief Title: Ga-68 Prostate Specific Membrane Antigen PET/CT in Gliomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Girish Kumar Parida, Assistant Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T/IMF/21/22/04
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Glioma; Astrocytoma; Anaplastic Astrocytoma; Oligodendroglioma; Glioblastoma Multiforme
Keywords: FDG PET-CT; PSMA PET-CT; MRI brain; Glioma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficiency of 68 Ga-PSMA-11 PET-CT in detection of recurrent gliomas (Experimental): Primary objective Detection of sensitivity and specificity of 68Ga PSMA-11 PET-CT to diagnose disease recurrence in gliomas Secondary objectives
  1. Comparison of tumor SUVmax between 68Ga-PSMA and 18F-FDG PET-CT images
  2. Comparison of sensitivity and specificity of Ga-68 PSMA-11 PET-CT with that of CEMRI in diagnosing disease recurrence in gliomas
  3. Correlation between WHO tumor grade in histology and SUVmax of the recurrent lesion on 68Ga- PSMA PET-CT scan
  4. Correlation between PSMA expression in histopathology specimen (using IHC) and SUVmax of recurrent lesion on 68Ga- PSMA PET-CT scan.
  5. Any adverse events of Ga-68 PSMA-11 will be recorded according to CTCAE
  Interventions: Diagnostic Test: PSMA PET-CT

INTERVENTIONS:
Diagnostic Test: PSMA PET-CT — Prostate Specific Membrane Antigen PET-CT

SUMMARY:
As a part of molecular imaging, many PET tracers have been investigated in this regard. Those include 18F-FDG being glucose analogue, 18F-FLT representing nucleoside metabolism, and 18F-FDOPA, 18F-FET, 11C-MET as amino acids analogues. Among these, 18F-FDG is the most commonly used tracer due to its broader use and easy availability. However, high physiological uptake in the brain is a significant limitation. The main limitation of other tracers is the need for onsite cyclotrons for their production, making their availability difficult. So, the search for an ideal modality is still ongoing, and the latest addition to this search is a radio ligand labeled Prostate Specific Membrane Antigen (PSMA). It is a new but potentially promising radiotracer, currently showing its utility in different malignancies. Investigators, therefore, aim to identify whether Ga-68 PSMA PET-CT has better diagnostic accuracy in the detection of recurrent gliomas than conventional imaging modalities.

DETAILED DESCRIPTION:
Prostate Specific Membrane Antigen (PSMA is a type II membrane glycoprotein and is typically overexpressed in primary and metastatic lesions of prostate malignancy as the name suggests. However, this overexpression is not limited to prostate cancer only. It has been reported that, PSMA is overtly expressed in the vascular endothelium of various other malignancies where significant neovascularization is seen. Gliomas being highly vascularized tumors, have shown significant PSMA expression in their vascular endothelium especially in high grade ones. If this PSMA expression can be assessed through noninvasive molecular imaging, this would further ease the management these tumors. Different lesions have shown different grades of PSMA uptake in the PET/CT with high grade gliomas showing high uptake. Most of the articles published till date are either case reports or studies comprising very few numbers of patients. We would like to use the PET tracer Ga -68 PSMA for the detection of recurrence in patients with glioma.

Investigators believe that 68 Ga PSMA PET-CT has the potential to play an imperative role in noninvasively evaluating recurrent gliomas and can overcome the limitations of the currently used modalities. Besides, extrapolation of the PSMA expression, which is indirect evidence of neovascularization, can also be used to assess treatment options like VEGF inhibitors (Bevacizumab). These studies can also pave the way for further studies involving PSMA-based radio ligand therapy, which is currently being successfully applied in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age more than18 years.
* Patients having past history of histologically proven glioma.
* Patients who have undergone prior treatment with tumor resection and/or radiation therapy and/or chemotherapy.
* Clinically suspected cases of recurrence.
* Patient should be willing to and able to give written informed consent

Exclusion Criteria:

* Pregnant lady.
* Breastfeeding mother.
* Patients who will deny to give consent.
* Any brain primary other than high grade glioma
* Patient diagnosed with other primary malignancy
* Patient with life threating neurological emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Detection of sensitivity and specificity of 68Ga PSMA-11 PET-CT to diagnose disease recurrence in gliomas | 3 months
  Detection of sensitivity and specificity of 68Ga PSMA-11 PET-CT to diagnose disease recurrence in gliomas

SECONDARY OUTCOMES:
Comparison of tumor SUVmax between 68Ga-PSMA and 18F-FDG PET-CT images | 3 months
  Comparison of tumor SUVmax between 68Ga-PSMA and 18F-FDG PET-CT images
Comparison of sensitivity and specificity of Ga-68 PSMA-11 PET-CT with that of CEMRI in diagnosing disease recurrence in gliomas | 3 months
  Comparison of sensitivity and specificity of Ga-68 PSMA-11 PET-CT with that of CEMRI in diagnosing disease recurrence in gliomas
Correlation between WHO tumor grade in histology and SUVmax of the recurrent lesion on 68Ga- PSMA PET-CT scan | 3 months
  Correlation between WHO tumor grade in histology and SUVmax of the recurrent lesion on 68Ga- PSMA PET-CT scan
Correlation between PSMA expression in histopathology specimen (using IHC) and SUVmax of recurrent lesion on 68Ga- PSMA PET-CT scan. | 3 months
  Correlation between PSMA expression in histopathology specimen (using IHC) and

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
IPD data will be shared after obtaining permission from the institute post completion of the study